CLINICAL TRIAL: NCT03736915
Title: A Trial Comparing Pain During Local Tumesent Injection In Fingers Using Different Syringe-Needle Combinations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 18-04-0421
Record Dates: First submitted 2018-06-24; First posted 2018-11-09 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Anesthesia, Local; Infiltration; Injection Site; Pain
Keywords: hand; injections; pain; syringes; anesthesia, local
MeSH Terms: conditions — Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: : A randomized single-blinded controlled trial is designed for 30 adult male healthy subjects to compare the pain from injection using syringe and needle combination i.e. 1) 1 cc syringe with 26G needle, 2) 3 cc syringe with 26 G needle, and 3) 5 cc needle with 26 G needle. The injection will be performed in any of at the second, third and fourth fingers of either subject's hand randomly. The injection will be SIMPLE block technique using 1 cc of NaCl 0.9% solution under the injection speed of 30 seconds/cc. Subjects are required to rate two check-point of VAS at the timing of needle puncture and just right after the completion of the infiltration. Upon the completion of each finger, the subject is also asked to give response to seri of questions regarding the procedures and their preferences. At the end of all injections, subject is asked to rate his preference of syringe and needle combination.
Who Masked: Participant, Outcomes Assessor
Masking Description: The senior author (T.O.H.P) will perform all injection, and are given three pieces of paper before ever injection, to silently give information on tumescent technique, fingers sequence, syringe-needle combinations sequence and the solution used. Subjects are seated comfortably, behind a screen with a small opening large enough to introduce the tested hand. Both hands are placed on the supine position on the table. Seating positions and hand positions are designed somewhat ergonomics and comfort, to avoid creating bias due to positional discomfort. They could not see any of the procedure and won't know which syringe-needle combinations is used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 cc syringe with 26 G needle (Active Comparator): comparing the pain from injection using syringe and needle combination i.e. 1) 1 cc syringe with 26G needle, 2) 3 cc syringe with 26 G needle, and 3) 5 cc needle with 26 G needle. The injection will be performed in any of at the second, third and fourth fingers of either subject's hand randomly. Injection using 1 cc of NaCl 0.9% solution under the injection speed of 30 seconds/cc.
  Interventions: Procedure: Injection using 1 cc of NaCl 0.9%; Other: Patient Preference Question; Other: Questionnaires
- 3 cc syringe with 26 G needle (Active Comparator): comparing the pain from injection using syringe and needle combination i.e. 1) 1 cc syringe with 26G needle, 2) 3 cc syringe with 26 G needle, and 3) 5 cc needle with 26 G needle. The injection will be performed in any of at the second, third and fourth fingers of either subject's hand randomly. Injection using 1 cc of NaCl 0.9% solution under the injection speed of 30 seconds/cc.
  Interventions: Procedure: Injection using 1 cc of NaCl 0.9%; Other: Patient Preference Question; Other: Questionnaires
- 5 cc needle with 26 G needle (Active Comparator): comparing the pain from injection using syringe and needle combination i.e. 1) 1 cc syringe with 26G needle, 2) 3 cc syringe with 26 G needle, and 3) 5 cc needle with 26 G needle. The injection will be performed in any of at the second, third and fourth fingers of either subject's hand randomly. Injection using 1 cc of NaCl 0.9% solution under the injection speed of 30 seconds/cc.
  Interventions: Procedure: Injection using 1 cc of NaCl 0.9%; Other: Patient Preference Question; Other: Questionnaires

INTERVENTIONS:
Procedure: Injection using 1 cc of NaCl 0.9% — The injection will be using SIMPLE block technique using 1 cc of NaCl 0.9% solution under the injection speed of 30 seconds/cc.
Other: Patient Preference Question — Patient is asked at the end of each injection which injection they prefer
Other: Questionnaires — Patient is asked to answer questionairres at the end of each injection

SUMMARY:
Background: This study aims to obtain the most favorable syringe and needle combination, which causes the least pain during local anesthesia tumescent injection in the simulation of fully awake hand surgery.

Methods: A randomized single-blinded controlled trial is designed for 30 adult male healthy subjects to compare the pain from injection using syringe and needle combination i.e. 1) 1 cc syringe with 26G needle, 2) 3 cc syringe with 26 G needle, and 3) 5 cc needle with 26 G needle. The injection will be performed in any of at the second, third and fourth fingers of either subject's hand randomly. The injection will be SIMPLE block technique using 1 cc of NaCl 0.9% solution under the injection speed of 30 seconds/cc. Subjects are required to rate two check-point of VAS at the timing of needle puncture and just right after the completion of the infiltration. Upon the completion of each finger, the subject is also asked to give response to seri of questions regarding the procedures and their preferences. At the end of all injections, subject is asked to rate his preference of syringe and needle combination.

DETAILED DESCRIPTION:
METHODS

3.1 DESIGN This is a randomized, single-blinded controlled trial to measure local pain following local anesthesia tumescent injection using a different combination of syringe and needle in a healthy volunteer.

3.2 TIME AND PLACE The study will be conducted at Cipto Mangunkusumo Hospital (RSCM) in February to March 2018

3.3 SAMPLE 30 male healthy subjects (aged 18-60 years) who volunteer to join this study and meet the inclusion criteria are going to be selected with the convenient sampling method

3.4 SAMPLE SIZE Sample size for pilot study are used. The expected sample size is between 10-40 per groups, therefore we choose 30 subjects (90 fingers tested) to be included into 3 different treatment group

3.5 INCLUSION AND EXCLUSION CRITERIA As for the trial, we will include subjects who are healthy in general, male and aged 18 to 60 years old. However, we also plan to exclude subjects with history of blood or coagulation disorder, history of neuro vasculopathy, history of liver and renal disease, currently active smoker or already stopped less than 1 month, had previous injury or surgery in hand, or hand scar detected, history of Raynaud's phenomenon, history of vasospastic disorders, history of scleroderma, history of Buerger's disease, history of Dupuytren's disease, and history of complex regional pain syndrome.

3.6 SUBJECTS ENROLLMENT Sampling method used are convenient method

3.7 METHODS Healthy subjects who met the inclusion criteria are included in the study. Subjects are given explanations about the research and are requested to sign the informed consent form, should they agree to join the study. Each subject will be assigned to three injections using different combination of syringe and needle: 1. 1 cc syringe with 26 G needle, 2. 3 cc syringe with 26 G needle and 3. 5 cc needle with 26 G needle. The injection will be randomized to take place in any of at the second, third and fourth fingers of both hands. Once one side is injected, the subject is asked to introduce the second hand, and for the third injection, the hand is changed again. No washout periods are intentionally given between needles.

Every subject is randomized into treatment of sequence using digital random generator from www.randomizer.org. The first sequence for randomization is syringe choice, (code 1cc =1, 3 cc= 2., 5cc=3) randomized for 30 sets, with no repetition. The second sequence for randomization is the hand choice (left hand=1, right hand=2) randomized for 30 sets, with repetition. The third sequence for randomization is the finger choice for either hand (2nd finger=1, 3rd finger=2, 4th finger=3) randomized for 30 sets, with repetition. The example for subject randomization table are shown at APPENDICES.

The injection technique used is SIMPLE block. A SIMPLE block is a block technique using infiltration where the point of needle injection is at the digitopalmar crease at its mid-axis. The tumescent solution used is Normal Saline (NaCl 0.9%), the amount of solution is one cc for each finger. We do not use lidocaine or anesthetic agents to avoid the bias of reduced pain along the course of injection. The rates of injection of each finger are 30 seconds (slow infusion) to inject all one cc of tumescent solution subcutaneously, regardless of syringe-needle combinations used. The metronome with the rate of 120 BPM is used so that the injection rate is constant along 30 s period. The metronome was used using headphone in injector ear, to avoid bias and creating anxiety to the subjects. The senior author (T.O.H.P) will perform all injection, and are given three pieces of paper before ever injection, to silently give information on tumescent technique, fingers sequence, syringe-needle combinations sequence and the solution used. Subjects are seated comfortably, behind a screen with a small opening large enough to introduce the tested hand. Both hands are placed on the supine position on the table. Seating positions and hand positions are designed somewhat ergonomics and comfort, to avoid creating bias due to positional discomfort. They could not see any of the procedure and won't know which syringe-needle combinations is used. The ambiance of procedure's room is situated to be silent, no music or unnecessary sounds are made. Subjects are actively communicated of what treatment is coming next during the procedures, so the readiness of subjects is precipitated.

A baseline subjective pain was marked by the subject using VAS, with the pain score from 1-10, 1 (very mild pain) to 10 (worst pain ever). VAS chart along with description placed on the table within subject's visual field. Pen are prepared so the subjects could mark their VAS score on the chart, with non-injected hand, when asked by operator. Its ensured that operator don't know the score when VAS noted to avoid bias. The person in charge of randomization prepared the syringe-needle combinations and solution as stated in the envelope. He/she also note the VAS score during all the injection and distribute the questionnaire after each injection.

The region of injection was sterilized with 70 % alcohol, and a waiting duration of 30 s was provided for total evaporation. The point needle insertion is at digitopalmar crease at its mid-axis at selected fingers. The procedure initiated by pinching the needle insertion point using operator fingers to create the tactile distraction, pinching is maintained for 10 seconds. Then the needle inserted in a perpendicular fashion (90 degrees to the skin surface), needles are proceeded down subcutaneously just beneath the dermis. Patient is asked the VAS score at this point (Check-point 1-needle prick). After the needles inserted subcutaneously, 30 second period of waiting is given to let the patient adapt to the needle prick pain. After 30 seconds, the infiltration of the tumescent solution is initiated. All one cc of the tumescent solution is infiltrated into the tissues within 30 seconds regardless of the syringe size, metronome with 120 bpm are used to control the rate. Two check-point of VAS are noted: the first initial injection and just after the completion of the infiltration. For all injections, the needle was kept subcutaneous for whole procedures with great care to stand still and minimize movement. Fresh needles are used when moving from one finger to the other fingers.

Upon the completion of each fingers, the subject is asked to give answer to series of a question regarding the procedures and their preferences. The answer given is written by giving only checks or cross on the question papers, so that patient can use any hand to write the answer with ease. Thus, these moments also could give some washout period for pain from the injected hand before. At the end of all injections, subjects are asked which combinations of syringe and needle they are preferred. The subjects were provided with four tablets of paracetamol 500 mg after the whole injection for they to take in case he suffers persistent pain. Subjects are asked to contact the researchers if pain persists or any adverse event occurred.

Some parameters, which will be recorded and documented are: 1. Pain scale using VAS during three checkpoints which are initial needle prick, initial infiltration of tumescent injection and after the infiltration finished, 2. Patient responses and preference regarding the procedures using questionnaire and 3. Patient preference of combinations of syringe and needle

3.8 VARIABLE The research design includes several independent variables to be tested such as: 1 cc syringe with 26 G needle, 3 cc syringe with 26 G needle and 5 cc needle with 26 G needle, tumescent solution used which is 1 cc NaCl 0.9% and finally the 3 choices of finger to be injected which are selected between 2nd, 3rd or 4th finger on both hands. The dependent variable in this study that will be analyzed are VAS score during three checkpoints; the initial needle prick, the initial infiltration of tumescent injection, and after all the infiltration finished, the patient preference and responses in patient preference questionnaire are also tested, along with the patient choices of injections kits.

3.9 OPERATIONAL DEFINITION

* 2nd finger: index finger in either hand
* 3rd finger: long finger in either hand
* 4th finger: ring finger in either hand
* SIMPLE finger block is a block technique using infiltration where the point of needle injection is at the digitopalmar crease at its mid-axis.
* Tumescent solution: The solution injected to finger during anesthesia, here we use Normal Saline (NaCl 0.9%) only. The amount of solution is 1 cc for each finger.
* Rates of injection: the speed or time required to inject all solution in the syringe to fingers
* The Visual Analogue Scale (VAS) a subjective measure of pain that consist of a 10-cm line with two end-point representing "no pain" and "worst pain imaginable." Subjects were asked to rate their pain by placing mark on the line corresponding to their current level of pain. The length along the line from "no pain" marker was then measured with a ruler giving a pain score out of 10. The VAS chart is translated into Bahasa Indonesia.
* 1 cc syringe: in this research, we are using 1 cc syringe produced by Terumo® (Terumo Corporation; Tokyo, Japan)
* 3 cc syringe: in this research, we are using 3 cc syringe produced by Terumo®
* 5 cc syringe: in this research, we are using 5 cc syringe produced by Terumo®
* 26-gauge needle: in this research, we are using 27-gauge needle produced by Terumo®
* Questionnaire: series of questionnaire asked after each injection procedure to assess patient preferences and responses. The questionnaire is translated into Bahasa Indonesia.

3.10 DATA ANALYSIS In this research, data processing is performed using an SPSS version 22.0 software. We assume that variance for each finger injected is the same (no significance difference). For VAS score data is presented a table and graphic form of the mean and standard deviation for numerical data, and with normal distribution and median. Minimum and maximum for numerical data with abnormal distribution. An ANOVA test analysis were used if the distribution is normal, Kruskall Wallis test analysis is used if the distribution is not normal, to assess the significance of three combinations of syringe and needle and VAS. The response for questionnaire also analyzed for their correlation with syringe used using chi square test. The significance level was set at P<0.05 with Confidence Interval 95%.

ELIGIBILITY:
Inclusion Criteria:

* healthy in general
* male sex
* aged 18 to 60 years old

Exclusion Criteria:

* history of blood or coagulation disorder
* history of neuro vasculopathy
* history of liver and renal disease
* currently active smoker or already stopped less than 1 month
* had previous injury or surgery in hand
* hand scar detected
* history of Raynaud's phenomenon
* history of vasospastic disorders
* history of scleroderma
* history of Buerger's disease
* history of Dupuytren's disease
* history of complex regional pain syndrome.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male biological sex
Enrollment: 30 (Estimated)
Dates: Start 2018-11-14 (Actual); Primary Completion 2018-11-19 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Pain measured using Visual Analagoue Scale (VAS) | VAS will be assessed at 3 check point: 1.Initial needle prick, 2.initial infiltration of tumescent injection and 3. after the infiltration finished
  VAS is usually a horizontal line using a 10 cm baseline, anchored by word descriptors at each end. The client is asked to mark a point on a continous line corresponding to the severity of their pain (from the left-end to right end range is from "no pain" to "pain as bad as it could possibly be")

SECONDARY OUTCOMES:
Patient questionnaire responses | Right after all injection sequence performed in one finger (approximately 10 seconds after the injection)
  Patient responses and preference regarding the procedures using 5 question with multiple choice questionnaire
Patient preference questionnaire | Right after all injection performed (approximately 50 seconds after all injection finished)
  Patient preference on which the injection procedures they prefer, using 1 question with multiple choice questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Theddeus Prasetyono, M.D., Principal Investigator — Division of Plastic Surgery, Faculty of Medicine University of Indonesia
Locations (1):
- ICTEC - Ciptomangunkusumo National Hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided